CLINICAL TRIAL: NCT06509256
Title: Different Methods of Tranexamic Acid Application in Controlling Perio Operative Bleeding in Gynecomastia
Brief Title: Different Methods of Tranexamic Acid Application in Controlling Peri Operative Bleeding in Gynecomastia Surgery
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amjad Ahmed Qasim AL-Gubari, Resident of Plastic Surgery, Department of Plastic and Reconstructive Surgery, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: plastic surgery department
Record Dates: First submitted 2024-06-08; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pharmacological-Aggravated Urticaria
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tumescent solution only (Control group) (Active Comparator): "The operative site will be injected with a standard tumescent solution prepared by adding 20ml of 2% lignocaine and 1ml of 1 in 1000 adrenaline to 500 ml of ringer lactate. No tranexamic acid will be used in this group."
  - All patients will undergo suction-assisted liposuction through an infra-areolar incision, followed by glandular excision using the orange peel excision technique. The surgical intervention will be performed as a day-care procedure. Patients will wear pressure garments continuously for 3 days post-operatively and intermittently and by the 3rd day we estimate the ecchymosis in the chest area then pressure garment will be reapplied for 7 to 10 days. Follow-up evaluations will be conducted immediately post-op, at 10 days.
  Interventions: Drug: Tranexamic acid injection
- Tumescent solution with tranexamic acid added (Active Comparator): "The operative site will be injected with a tumescent solution prepared as in Group A (Control group), with the addition of 500 mg tranexamic acid to the tumescent solution."
  - All patients will undergo suction-assisted liposuction through an infra-areolar incision, followed by glandular excision using the orange peel excision technique. The surgical intervention will be performed as a day-care procedure. Patients will wear pressure garments continuously for 3 days post-operatively and intermittently and by the 3rd day we estimate the ecchymosis in the chest area then pressure garment will be reapplied for 7 to 10 days. Follow-up evaluations will be conducted immediately post-op, at 10 days.
  Interventions: Drug: Tranexamic acid injection
- Tumescent solution with intravenous tranexamic acid (Active Comparator): The standard tumescent solution as in the control group, with 500 mg tranexamic acid administered intravenously ( well-injected IV directly).
  - All patients will undergo suction-assisted liposuction through an infra-areolar incision, followed by glandular excision using the orange peel excision technique. The surgical intervention will be performed as a day-care procedure. Patients will wear pressure garments continuously for 3 days post-operatively and intermittently and by the 3rd day we estimate the ecchymosis in the chest area then pressure garment will be reapplied for 7 to 10 days. Follow-up evaluations will be conducted immediately post-op, at 10 days.
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — work aims to evaluate the role of tranexamic acid in bleeding control in gynecomastia surgery

SUMMARY:
Different Methods of Tranexamic Acid Application in Controlling Peri-Operative Bleeding in Gynecomastia Surgery

DETAILED DESCRIPTION:
The term "gynecomastia" is derived from the Greek words "gyne" = woman and "mastos" = breast and is a benign enlargement of the male breast. It is the most common condition affecting the male breast due to enlargement of both ductal and stromal tissue[1].

Plastic surgeons frequently perform gynecomastia operations as cosmetic procedures. Since these operations result in relatively little blood loss, there is little information in the literature about how to minimise blood loss during these cosmetic procedures Some preventive measure against bleeding and hematomas include perioperative blood pressure control, use compressive dressing, different types of suction drains, size of incision, careful hemostasis, and infusion of adrenalin during local anesthesia, infusion of tranexamic acid in tumescent or intravenous directly

ELIGIBILITY:
Inclusion Criteria:

* Age (16 - 45 years)
* Any grade of gynecomastia well be included

Exclusion Criteria:

* Age (<16 - >40 years)
* History of previous gynecomastia surgery
* Patients with known allergy to tranexamic acid
* Patients with abnormal coagulation profile (according to American Society of Anesthesiologists guidelines for preoperative preparation of surgical patients)
* Patients who are receiving treatment for known hyper-coagulable state. 6. Patients with history of cardiac disease or thromboembolic events.

Ages: 16 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss during liposuction in milliliters | "Intraoperatively" Unit of Measure: Milliliters (mL)
  The volume of blood collected in the liposuction bottle during the surgical procedure will be measured. This will be reported as mean volume in milliliters with standard deviation for each study group.

SECONDARY OUTCOMES:
Duration of surgical drain placement in days | From immediate post-operation until drain removal (expected within 3 to 7 days)" Unit of Measure: Days
  The number of days the surgical drain remains in place post-operatively, until drainage is less than 30 mL per 24 hours. This will be reported as mean number of days with standard deviation for each study group.
Change in hemoglobin concentration from baseline to 24 hours post-operation | Baseline (within 24 hours before surgery) and 24 hours post-operation" Unit of Measure: Grams per deciliter (g/dL)
  The difference in hemoglobin concentration between preoperative baseline and 24 hours post-operation. This will be reported as mean change in g/dL with standard deviation for each study group.
Extent of post-operative ecchymosis at 7 days | "7 days post-operation" Unit of Measure: Ordinal scale score (0-4)
  The extent of ecchymosis will be assessed using a standardized photographic scale, ranging from 0 (no ecchymosis) to 4 (severe ecchymosis). This will be reported as median score with interquartile range for each study group."
Changes in coagulation profile at 24 hours post-operation | "Baseline (within 24 hours before surgery) and 24 hours post-operation" Unit of Measure: Seconds for PT and aPTT, no units for INR
  Changes in prothrombin time (PT), activated partial thromboplastin time (aPTT), and international normalized ratio (INR) from baseline to 24 hours post-operation. These will be reported as mean changes with standard deviations for each parameter in each study group.

IPD SHARING:
Plan to Share IPD: Yes